CLINICAL TRIAL: NCT07078435
Title: Inflammation, Innate Immunity, MIcrobiota and Inovative Treatments in ENDOmetriosis
Brief Title: Innate Immunity, MIcrobiota and Inovative Treatments in Endometriosis
Acronym: IMIEndo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC25.0052
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis; Immunity; Microbiota
Keywords: endometriosis; surgery; immunity; efferocytose; microbiota
MeSH Terms: conditions — Endometriosis | interventions — Surgical Procedures, Operative; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: This study is a monocentric (at Grenoble University Hospital), open-label, prospective experimental study with a control arm.
  Given the extent of the biopsies performed during surgery, which exceed standard care, French legislation classifies this study as a Class 2 interventional study.
  Women in the endometriosis group will undergo collection during surgery with endometriotic lesions, adjacent tissue, eutopic endometrium, and peritoneal lavage during surgery. Controls will provide biopsies of eutopic endometrium, unaffected peritoneum, and peritoneal lavage during the gynecology surgery.
  For both groups, peripheral blood samples will be collected during routine care and stool samples obtained. For the endometriosis group, a second stool sample will be collected at 12 months.
  A clinical evaluation will be performed at inclusion for all participants and repeated at one year for the endometriosis group. Participation for control group subjects is limited to the day of surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometriosis group (Active Comparator): Patients in "endometriosis group" are aged 18-42 years and suffer symptomatic endometriosis that requires a surgery indication (due to persistent symptoms despite medical treatment and/or risk of organ damage). These patients generally undergo hormonal therapy, but this must be discontinued at least one month prior to surgery. The surgery is scheduled to take place during the luteal phase.
  Patients don't take a immunosuppressor, antibiotic or present inflammatory bowel disease, recent infection, pregnancy
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines; Biological: Blood test; Biological: Stool samples
- Control group (Active Comparator): Patients in "control group" are aged 18-42 years and don't suffer endometriosis that requires a gynecological surgery indication (permanent contraception, benine surgery). The surgery is scheduled to take place during the luteal phase. Patients don't take a immunosuppressor, antibiotic or present inflammatory bowel disease, recent infection, pregnancy
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines; Biological: Blood test; Biological: Stool samples

INTERVENTIONS:
Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — The surgery is performed on both arms as part of the current / recommended treatment. But during this surgery, an extension of the samples is performed. In both arms, the surgeons take samples of the endometrium, peritoneum and peritoneal lavage. For patients with endometriosis, the lesion is also sampled.
Biological: Blood test — Before surgery, the patient will need a blood test at the recommendation of the anaesthetist. This allows us to see the level of oestrogen and progesterone in the blood.
Biological: Stool samples — Before the surgery, the patient will take a stool sample.
Biological: Stool samples — After 1 year's follow-up, the patient will take a stool sample.
  Arms: Endometriosis group

SUMMARY:
Endometriosis is a chronic inflammatory, polygenic, and multifactorial disease affecting approximately 10% of women of reproductive age, corresponding to over one million women in France. Endometriosis profoundly impairs the health and quality of life of affected individuals and carries a significant socio-economic burden, making it a major public health concern. To date, the pathogenesis and prognostic factors of disease progression remain poorly understood. Despite current treatment options, which are based on hormonal therapy or surgery, resistance and recurrence are frequent, underscoring the urgent need for innovative therapeutic strategies.

The hypothesis of retrograde menstruation of endometrial cells, among other proposed theories, appears insufficient to fully explain the development of the disease. Immunological factors may be implicated. Endometriosis is characterized by the presence of endometriotic tissue outside the uterine cavity- within the peritoneal cavity or at distant sites-forming lesions that, like eutopic endometrium, contain infiltrating immune cells, with varying compositions across menstrual cycle phases. Although data remain scarce, the literature points to several key mechanisms:

Inflammation and innate immunity with the dendritic cells, that initiate and orchestrate immune responses, appear to be present in different proportions and exhibit altered phenotypes in endometriotic tissue compared to healthy tissue. Macrophages, essential for phagocytosis, tissue repair, and the resolution of inflammation, also show functional and phenotypic modulation. In particular, efferocytosis-their ability to clear apoptotic cells-is impaired, and an imbalance in M1/M2 polarization has been described, potentially facilitating menstrual cell escape. The local microenvironment is characterized by altered cytokine and chemokine profiles. Natural Killer cells exhibit disrupted expression patterns of activating and degranulation capacity.

Microbiota: Many studies suggest a potential role for the intestinal microbiota in the initiation and/or promotion of endometriosis. Patients frequently exhibit gut dysbiosis, marked by reduced microbial diversity.

Resolution of Inflammation: Endometriosis may be associated with defective resolution of inflammation. Resolutive pharmacology involves the use of pro-resolving factors to exert a therapeutic effect by accelerating or stimulating the resolution of inflammation.

The interplay between local inflammation, the gut microbiota, and disease progression remains incompletely elucidated. A comprehensive phenotypic and functional characterization of immune cells-particularly innate immune cells (dendritic cells, macrophages, Natural Killer cells) - in parallel with microbiome profiling and clinical outcome data, may yield novel insights into disease mechanisms and support the development of pro-resolutive therapeutic strategies that may be of interest in endometriosis.

Study Design This will be a monocentric (at Grenoble University Hospital), open-label, prospective experimental study with a control arm.

The primary objective is to identify immune biomarkers associated with endometriosis.

Secondary objectives include:

1. Identification of immune biomarkers associated with clinical outcomes in endometriosis.
2. Characterization of the immunogenetic KIR/HLA (Killer Immunoglobulin-like Receptors / Human Leukocyte Antigen) system in both study groups.
3. Analysis of stromal cells, apoptosis, macrophage efferocytosis, and their responsiveness to pro-resolutive factors in both groups.
4. Identification of a characteristic bacterial gut microbiota profile at diagnosis in women with endometriosis versus controls, and/or profiles associated with one-year clinical outcomes (favorable vs unfavorable), as well as temporal microbiota trajectories over one year in relation to clinical response.

Study Population:

The study will include women undergoing surgery for endometriosis versus control women undergoing benign gynecological surgery with no known history or intraoperative evidence of endometriosis, aged 18 to 42.

Study Procedures:

Women in the endometriosis group will undergo collection of endometriotic lesions, adjacent tissue, eutopic endometrium, and peritoneal lavage during surgery. Controls will provide biopsies of eutopic endometrium, unaffected peritoneum, and peritoneal lavage. For both groups, peripheral blood samples will be collected during routine care and stool samples obtained at baseline (Day 0). For the endometriosis group, a second stool sample will be collected at 12 months (M12).

A clinical evaluation will be performed at inclusion for all participants and repeated at one year for the endometriosis group. Participation for control group subjects is limited to the day of surgery, whereas endometriosis group subjects will be followed for 12 months.

DETAILED DESCRIPTION:
Introduction Endometriosis is a chronic inflammatory, polygenic, and multifactorial disease affecting approximately 10% of women of reproductive age, corresponding to over one million women in France. Endometriosis profoundly impairs the health and quality of life of affected individuals and carries a significant socio-economic burden, making it a major public health concern. To date, the pathogenesis and prognostic factors of disease progression remain poorly understood. Despite current treatment options, which are based on hormonal therapy or surgery, resistance and recurrence are frequent, underscoring the urgent need for innovative therapeutic strategies.

The hypothesis of retrograde menstruation of endometrial cells, among other proposed theories, appears insufficient to fully explain the development of the disease. Immunological factors may be implicated. Endometriosis is characterized by the presence of endometriotic tissue outside the uterine cavity - within the peritoneal cavity or at distant sites - forming lesions that, like eutopic endometrium, contain infiltrating immune cells, with varying compositions across menstrual cycle phases. Although few data remain, the literature points to several key mechanisms:

Inflammation and Innate Immunity: Dendritic cells (DC), pivotal in initiating and orchestrating immune responses, appear to be present in different proportions and exhibit altered phenotypes in endometriotic tissue compared to healthy tissue. Macrophages, essential for phagocytosis, tissue repair, and the resolution of inflammation, also show functional and phenotypic modulation. In particular, efferocytosis-their ability to clear apoptotic cells-is impaired, and an imbalance in M1/M2 polarization has been described, potentially facilitating menstrual cell escape. The local microenvironment is characterized by altered cytokine and chemokine profiles, with interleukin-8 (IL-8) potentially playing a key role via its angiogenic and chemoattractant properties. Natural Killer (NK) cells exhibit disrupted expression patterns of activating and inhibitory Killer-cell Immunoglobulin-like Receptors (KIRs), alongside diminished IFN - gamma (InterFeroN) secretion and degranulation capacity.

Microbiota: It is now well established that the immune system maintains a dynamic interaction with the gut microbiota at the mucosal barrier, with reciprocal modulation of local and systemic immunity. Furthermore, endometriosis is a hormone-sensitive pathology, and it is noteworthy that microbiota could increase plasma estrogen levels via β-glucuronidase-expressing bacteria. Other link with the microbiota, in mice, the treatment with antibiotics decrease the pathology. It is now well known that the dysbiosis can lead to systemic inflammation and subsequently contribute to inflammatory diseases development. A limited number of studies suggest a potential role for the intestinal microbiota in the initiation and/or promotion of endometriosis. Patients frequently exhibit gut dysbiosis, marked by reduced microbial diversity and an altered Firmicutes/Bacteroidetes ratio.

Resolution of Inflammation: Endometriosis may be associated with defective resolution of inflammation. Resolutive pharmacology involves the use of pro-resolving factors to exert a therapeutic effect by accelerating or stimulating the resolution of inflammation.

The biotechnology company Med'Inn'Pharma has developed a complex pro-resolving biological drug consisting of a macrophage supernatant that has eliminated apoptotic cells. This drug candidate has been used effectively in various experimental models of unresolved chronic inflammatory diseases, such as rheumatoid arthritis, multiple sclerosis and inflammatory bowel disease. In collagen-induced arthritis (a relevant model for rheumatoid arthritis), this drug candidate induces the reprogramming of macrophages towards a pro-resolving profile. The same applies to dendritic cells, with a significant reduction in the expression of costimulatory molecules.

The interplay between local inflammation, the gut microbiota, and disease progression remains incompletely elucidated. A comprehensive phenotypic and functional characterization of immune cells-particularly innate immune cells (dendritic cells, macrophages, NK cells)-in parallel with microbiome profiling and clinical outcome data, may yield novel insights into disease mechanisms and support the development of pro-resolutive therapeutic strategies.

Study Design This will be a monocentric (at Grenoble University Hospital), open-label, prospective experimental study with a control arm.

The primary objective is to identify immune biomarkers associated with endometriosis. The primary endpoint is the characterization and comparison of innate immune cells (both tissue-resident and circulating) across different biological compartments (blood, peritoneal fluid, biopsies), and between women with and without endometriosis ("endometriosis" vs "control" groups).

For that, we will perform immunophenotyping using flow cytometry on cells from each tissue (blood, endometrium, peritoneum, peritoneal lavage, and, for the endometriosis group, endometriotic lesions). A panel of approximately twenty fluorochrome-conjugated antibodies will be used to characterize the phenotype and activation status of each cell type within each tissue, including dendritic cells, macrophages, natural killer cells, and other innate immune cells. Cellular functionality will also be assessed by analyzing culture supernatants using the Luminex technique.

Secondary objectives include:

1. Identification of immune biomarkers associated with clinical outcomes in endometriosis.
2. Characterization of the immunogenetic KIR/HLA (Human Leukocyte Antigen) system in both study groups.
3. Analysis of stromal cells, apoptosis, macrophage efferocytosis, and their responsiveness to pro-resolutive factors in both groups.
4. Identification of a characteristic bacterial gut microbiota profile at diagnosis in women with endometriosis versus controls, and/or profiles associated with one-year clinical outcomes (favorable vs unfavorable), as well as temporal microbiota trajectories over one year in relation to clinical response.

Secondary endpoints include:

1. Description and comparison of innate immune cell populations (tissue and circulating) based on one-year clinical outcome (favorable vs unfavorable).

Immunogenetic profiling of HLA-A, -B, -C and KIR alleles by Next-Generation Sequencing (NGS), compared between women with and without endometriosis.

Stromal cell analysis:

* Comparison of stromal cell phenotypes, susceptibility to apoptosis, and macrophage efferocytosis capacity (using monocyte-derived macrophages) between cases and controls.
* Assessment of pro-resolutive factors' impact on macrophage efferocytosis.

Gut microbiota profiling:

Comparison of microbial community composition using 16S rDNA sequencing (relative abundances, Shannon and Bray-Curtis indices), and its evolution at 12 months (cases only), in relation to the presence of endometriosis and clinical outcome at one year.

Study Population:

The study will include women undergoing surgery for endometriosis versus control women undergoing benign gynecological surgery with no known history or intraoperative evidence of endometriosis. Patients should be young (18 to 42 years old) to ensure that, unfortunately, they may have endometriosis with predominantly inflammatory rather than fibrotic lesions. Furthermore, patients must not be undergoing immune modulation with antibiotics or immunosuppressive agents for the purposes of the study.

Study Procedures:

Women in the endometriosis group will undergo collection of endometriotic lesions, adjacent tissue, eutopic endometrium, and peritoneal lavage during surgery. Controls will provide biopsies of eutopic endometrium, unaffected peritoneum, and peritoneal lavage. These samples are collected by a gynecologic surgeon specialized in endometriosis.

For both groups, peripheral blood samples will be collected during routine care by the nurse and self stool samples obtained at baseline (Day 0). For the endometriosis group, a second stool sample will be collected at 12 months (M12).

No investigational treatment will be administered. But given the extent of biopsies performed during surgery, French legislation classifies this study as a Class 2 interventional study. The study has been approved by an ethics committee in accordance with French regulatory requirements.

A clinical evaluation will be performed at inclusion for all participants and repeated at one year for the endometriosis group. Participation for control group subjects is limited to the day of surgery, whereas endometriosis group subjects will be followed for 12 months.

The clinical evaluation focus on the medical history, the pain, the treatment. She is realized by surgeon.

All biological samples (blood, biopsies, peritoneal lavage, stool) will be processed and stored (plasma, cells, DNA, tissue) in a dedicated biobank for subsequent analysis. All samples will be collected at CHUGA.

Statistical Analysis

Given the expected sample size, appropriate non-parametric tests will be used. For each group, qualitative variables will be expressed as counts and percentages, and quantitative variables as mean ± standard deviation or median with interquartile range depending on the distribution. Comparisons will be conducted using Friedman, Wilcoxon, Mann-Whitney, or Student's t-tests, depending on data distribution, number of groups, and pairing status. Log-transformation will be applied if normality is not met. Primary comparisons will focus on immune cell parameters across tissues and study groups, including:

* Frequencies of immune cell subsets,
* Activation/maturation status,
* TLR ligand responses,
* KIR/HLA genotype combinations,
* Stromal cell apoptosis,
* Macrophage efferocytosis capacity,
* Gut microbiota composition (α-diversity: Shannon and Simpson indices; β-diversity: Bray-Curtis dissimilarity).

To control for multiple comparisons, Bonferroni correction may be applied. This exploratory study aims to identify candidate biomarkers and immunological signatures associated with endometriosis and disease recurrence, thereby generating hypotheses for future investigations.

Conclusion Endometriosis imposes a substantial burden on affected women and society. While no direct benefit is anticipated for participants, this study aims to advance the understanding of biological-especially immunological-mechanisms underpinning the disease. The results may support the identification of novel therapeutic targets, including agents that promote inflammation resolution. This research will help define an immunological signature of endometriosis, establish links with the gut microbiota, and assess the preclinical efficacy of a pro-resolutive biologic compound as a potential disease-modifying therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-42 years.
* Surgery scheduled during the luteal phase.
* Written informed consent provided.

Additional inclusion criteria for the "endometriosis" group:

* Women with confirmed endometriosis and a surgical indication (due to persistent symptoms despite medical treatment and/or risk of organ damage).
* Hormonal therapy discontinued at least one month prior to surgery.
* Absence of isolated ovarian endometrioma.

Control group inclusion criteria:

- Women requiring benign gynecological surgery with no clinical or intraoperative evidence of endometriosis.

No inclusion criteria (both groups):

* Presence of inflammatory bowel disease (Crohn's disease, ulcerative colitis) or other autoimmune disorders (e.g., lupus, Sjögren's syndrome, antiphospholipid syndrome, rheumatoid arthritis, spondyloarthritis),
* Use of antibiotics within the month prior to surgery,
* Recent infection (<2 weeks),
* Ongoing treatment with biologics or immunosuppressants,
* Contraindication to surgery due to general condition or comorbidities,
* Hormonal therapy within the month prior to surgery,
* Abdominopelvic surgery involving peritoneal breach within the previous 6 months,
* Pregnancy or breastfeeding,
* Participation in another clinical study (RIPH 1 or 2).

Exclusion Criteria:

* Intraoperative impossibility to perform surgery due to local conditions with an unfavorable benefit-risk balance for the patient.
* Discovery of endometriosis during surgery in the control group.
* Use of biologics or immunosuppressants within the first year after inclusion in the endometriosis group.
* Antibiotic use in the month preceding the second stool sample (endometriosis group).

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As endometriosis only affects non-menopausal women, the study concerns women of childbearing age. As it's the inflammatory lesions of endometriosis we're interested in, we need young patients, so we're limiting the age range to 18 to 42.
Enrollment: 40 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
To identify immune biomarkers associated with endometriosis. | The day of inclusion with the sample during the surgery
  The primary endpoint is to describe and compare innate immune cells (with dendritic cells, macrophages, natural killers cells, lymphocytes) according to tissue (blood, peritoneal lavage, biopsies of endometrium and more or less endometriosis) and for each tissue according to the presence of endometriosis ("endometriosis" and "control" groups).
  The variables analyzed will be the frequencies of different subpopulations of dendritic cells (cDC1, cDC2, PDC, inflammatory DC), macrophages (M0, M1, M2), and effectors (NK, iNKT, lymphocytes T); as well as their level of maturity or activation, assessed by their expression of surface markers relevant.

SECONDARY OUTCOMES:
To identify immune biomarkers associated with clinical response in endometriosis | The samples are collected during the day of surgery
  This objective consist to understand the link of immunity with evolution of endométriosis.
  The aim is to secondary outcomes whether the frequency of immune cells, their distribution and also their degree of activation is predictive of the development of endometriosis after surgery.
  The clinic will be separating on two groups : good evolution and bad evolution (= stable clinic or decline of health status).
To characterize the KIR/HLA (Human Leukocyte Antigen) immunogenetic system in both "endometriosis" and "control" groups | The sample are collected the surgery day.
  KIR/HLA genotyping will be performed using DNA extracted from the cells of women in both groups. HLA typing will be carried out using the laboratory's routine NGS techniques, and KIR typing by multiplex PCR using primers specific to each KIR gene, using NGS KIR technologies developed in Christelle Retière's laboratory at the EFS/INSERM laboratory in Nantes.
To characterize stromal cells, their apoptosis. | The samples are collected during the surgery day
  The phenotype of frozen stromal cells will be characterized by CD45, CD10, CD29, CD44, CD73, with analysis of the expression of NK inhibitory molecules HLA-E, HLA-C and HLA-G. Expression of estrogen and progesterone receptors will also be measured by flow cytometry. The sensitivity of these stromal cells to apoptosis will also be measured (AnnV/7AAD labelling, expression of pro- and anti-apoptotic factors by flow cytometry), in kinetics, in order to detect any failure of this apoptosis, and correlate it with the presence of macrophages and dendritic cells in the tissues.
To characterize macrophage efferocytosis this their response to pro-resolving factors in both "endometriosis" and "control" groups. | The samples are collected during the surgery day
  Blood monocytes will be differentiated into macrophages by culture, and their capacity for efferocytosis (phagocytosis of apoptotic cells), as well as that of tissue macrophages, will be assessed. A standardized test for this function has been developed by Sylvain Perruche's laboratory in Besançon. The macrophage secretome from the different patient groups will be characterized by microarrays and functional testing,
To identify a profile of bacterial intestinal microbiota at diagnosis characteristic of "endometriosis" patients compared with "controls", and/or associated with clinical response at 1 year (favorable or unfavorable). | The stools samples are collected the surgery day in hospitalisation and at the one year of follow up.
  This objective consist to understand the link of microbiota and endométriosis and/or her evolution with clinic.
  The clinic will be separating on two groups : good evolution and bad evolution (= stable clinic) Genomic extraction will be carried out on the stools collected, followed by qRT-PCR (Polymerase Chain Reaction) to estimate the total quantity of bacteria present in the TIMC (Translational and Innovative Medicine and Complexity) laboratory. Metagenomic analysis (16S RNA (RiboNucleic Acids)) will be carried out to determine the different phyla (and species) and their relative proportions. qRT-PCR analysis will be used to quantify some of the bacteria identified as most relevant in discriminating patients with and without endometriosis. The following parameters describing diversity a (Shannon index and Simpson index), and b (Bray-Curtis index) will be determined and compared. Microbiota data will also be analyzed using unsupervised (PCA) and supervised (PLS-DA) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Chaperot, PhD, Study Director — Etablissement Français du Sang; Thierry Michy, Dortor, Principal Investigator — Centre Universitaire Grenoble Alpes
Locations (1):
- CHUGA, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: Yes